CLINICAL TRIAL: NCT02760927
Title: Assessment of AnchorFast Guard Oral Endotracheal Tube Fastener on Patients Intubated With Oral Endotracheal Tubes With Subglottic Suction
Brief Title: Assessment of a Oral Endotracheal Tube Fastener on Patients Intubated With Oral Endotracheal Tubes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study product will not be commercialized.
Sponsor: Hollister Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5799-I
Record Dates: First submitted 2016-04-18; First posted 2016-05-04 (Estimated); Results first posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-08

CONDITIONS: Respiratory Depression; Respiratory Failure; Ventilatory Depression
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endotracheal Tube Fastener (Experimental): The intervention administered is a revised commercially available endotracheal tube holder with a tract to accommodate a subglottic suction lumen of an oral endotracheal tube.
  Interventions: Device: Endotracheal Tube Fastener

INTERVENTIONS:
Device: Endotracheal Tube Fastener — The AnchorFast Guard oral endotracheal tube fastener provides a convenient means to hold an oral endotracheal tube securely in place without the use of adhesive tape. The oral endotracheal tube fastener allows repositioning of the tube in either direction along the track without removal of the device.
  Other Names: AnchorFast Guard Oral Endotracheal Tube Fastener

SUMMARY:
Assessment of AnchorFast Guard Oral Endotracheal Tube Fastener on Patients Intubated with Oral Endotracheal Tubes with Subglottic Suction

DETAILED DESCRIPTION:
Endotracheal intubation is the trans laryngeal placement of a tube into the trachea via the nose or mouth. Subglottic suctioning, during endotracheal tube securement, is important for mechanically-ventilated patients to allow for the clearance of secretions that may accumulate during intubation. This protocol examines an enhancement to the current AnchorFast Guard device in order for the device to hold a subglottic suctioning lumen in addition to the intubation tube.

ELIGIBILITY:
Inclusion Criteria:

* Is 18 years of age or older and requires oral tracheal intubation
* Has intact skin on application site
* Is qualified to participate in the opinion of the Investigator including the requirement for endotracheal tube with subglottic suction

Exclusion Criteria:

* Has an existing neck injury
* Has protruding upper teeth, is without teeth or is unable to wear upper dentures
* Has facial hair
* Has clinically significant skin damage, condition or disease on the application site which may contraindicate participation
* Has a known or stated allergy to adhesive bandages, or any of the product types being tested
* Uses of topical drugs, lotions, creams or oils on the application site
* Is participating in any clinical testing which may affect performance of this device
* AnchorFast Guard Oral Endotracheal Tube Fastener does not fit subject's face

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Newton, JD, Study Chair — Legacy Research Institute IRB
Locations (3):
- United States (3):
  - Legacy Mt Hood, Gresham, Oregon
  - Legacy Good Samaritan, Portland, Oregon
  - Legacy Salmon Creek Medical Center, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Endotracheal Tube Fastener
Started | 4
Completed | 3
Not Completed | 1
Not completed — Tube Slippage from Device | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat principles followed. All four subjects were included in the analysis
Arm/Group | Endotracheal Tube Fastener
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethic Heritage: White (not of Hispanic origin) | 3
  Race/Ethic Heritage: Asian or Pacific Islander | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants on Which Test Product Allowed for Proper Placement of the Subglottic Suction Lumen
Description: Assessed by the proportion of yes/no researcher responses
Time Frame: Typical wear time of endotracheal tube fastener up to one week
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Tube Fastener
Number analyzed (Participants) | 4
Participants | 4

2. Primary Outcome: Proportion of Participants on Which the Subglottic Suction Lumen Was Easy to Place Into the Tract With the Tube Protection Sleeve
Description: Assessed by the proportion of researcher responses that equal agree (4) plus strongly agree (5) on a five point scale that includes strongly disagree (1) disagree (2) and no opinion (3)
Time Frame: Typical wear time of endotracheal tube fastener up to one week
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Tube Fastener
Number analyzed (Participants) | 4
Participants
  Strongly Agree | Agree | 3
  Strongly Disagree | Disagree | No opinion | 1

3. Primary Outcome: Proportion of Participants on Which the Test Product Allowed the Subglottic Suction Lumen to Remain Within the Subglottic Suction Lumen Tract
Description: Assessed by the proportion of yes/no researcher responses
Time Frame: Typical wear time of endotracheal tube fastener up to one week
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Tube Fastener
Number analyzed (Participants) | 4
Participants
  Yes | 3
  No (Thick secretions) | 1

4. Primary Outcome: Proportion of Participants on Which the Test Product Protected the Subglottic Suction Lumen
Description: Assessed by the proportion of yes/no researcher responses
Time Frame: Typical wear time of endotracheal tube fastener up to one week
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Tube Fastener
Number analyzed (Participants) | 4
Participants
  Yes | 3
  No (Removed with thick secretions) | 1

5. Primary Outcome: Proportion of Participants on Which the Test Product Allowed for Effective Subglottic Suctioning
Description: Assessed by the proportion of yes/no researcher responses
Time Frame: Typical wear time of endotracheal tube fastener up to one week
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Tube Fastener
Number analyzed (Participants) | 4
Participants
  Yes | 3
  No (Thick secretions) | 1

ADVERSE EVENTS:
Arm/Group | Endotracheal Tube Fastener
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endotracheal Tube Fastener (N=4)
Device-associated tongue displacement (Product Issues) | 2 (2) — Device-associated tongue displacement

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results of the trial are the exclusive and sole property of the Sponsor, and the Sponsor has the right to publish the results of the trial. Publication of results or release by the PI of information obtained for the Sponsor requires previous written approval and authorization by the Sponsor.